CLINICAL TRIAL: NCT06203236
Title: Natriuresis-Guided Diuretic Therapy in Patients With Acute Heart Failure With Reduced Ejection Fraction and Chronic Kidney Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Hisham Mohammed Hasan, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Natriuresis-Guided Diuretics
Record Dates: First submitted 2023-11-22; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Acute Heart Failure; Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natriuresis-guided group (Active Comparator): Natriuresis-guided therapy group receiving diuretic therapy guided by natriuresis measurements.
  Interventions: Drug: Furosemide 20 MG; Other: diuretic therapy
- Control group (Active Comparator): Patients with matched age and sex as control group receiving diuretic therapy only.
  Interventions: Drug: Furosemide 20 MG; Other: diuretic therapy

INTERVENTIONS:
Drug: Furosemide 20 MG — 1. The median daily total dose of intravenous loop diuretic at the start of treatment will be 20 mg of furosemide.
  2. Monitoring of urinary sodium excretion (natriuresis) and diuresis will begin 2 hours after treatment initiation.
  Other Names: Lasix 20 MG
Other: diuretic therapy — diuretic therapy

SUMMARY:
To investigate the effectiveness and feasibility of natriuresis-guided diuretic therapy as a personalized approach to managing acute heart failure in patients with underlying chronic kidney disease and its effect on short term outcomes.

DETAILED DESCRIPTION:
Natriuresis-guided diuretic therapy represents a promising approach in managing the complex and challenging clinical scenario of patients with acute heart failure (AHF) . These patients present a unique set of therapeutic dilemmas as traditional diuretic use to relieve congestion in AHF can potentially exacerbate renal dysfunction in those with preexisting CKD . Natriuresis-guided therapy improve patient centered outcomes by adjusting diuretic treatment based on the measurement of urinary sodium excretion which is feasible and able to improve decongestion in AHF with volume overload .

Patients with both AHF and CKD often experience disrupted fluid dynamics, biochemically, it appears covertly as an abnormality in renal function and when progressive, is manifested by symptom exacerbation and worsening renal impairment during application of therapy to ameliorate such symptoms. The pathways leading to these distinct impairments involve not only hemodynamic deterioration but also neurohormonal, inflammatory, and intrinsic renal mechanisms that produce this syndrome .

Natriuresis-guided diuretic therapy, by focusing on the excretion of sodium in the urine. Natriuresis-guided diuretic therapy assesses sodium excretion in urine, offering a direct way to gauge diuretic effectiveness in managing fluid in heart failure (HF) patients. In HF, neurohormonal activation can cause resistance to loop diuretics, leading to persistent congestion. Urinary sodium (UNa) measurement, recommended by ESC guidelines, helps evaluate diuretic response. Early UNa assessment aligns with observational studies, but controlled trials are ongoing. Traditional metrics like weight loss have limitations. UNa assessment can assist diuretic therapy, but factors like fluid overload severity, timing of assessment, kidney disease, and diuretic type should be considered .

One of the primary advantages of natriuresis-guided therapy is its potential to tailor treatment strategies to individual patient responses. It recognizes that not all patients with AHF and CKD will respond to diuretics in the same way. Natriuretic response measured via the urinary sodium (UNa) concentration in a urine spot sample has gained popularity as a metric used for early assessment of diuretic response. In patients with chronic kidney disease admitted for AHF, assessment of intrinsic renal sodium avidity using a random UNa spot sample provides an opportunity to gain insights into decongestive and diuretic responses to IV diuretic drug administration .

The concept of natriuresis-guided therapy represents a departure from the conventional one-size-fits-all treatment model in acute heart failure (AHF) management. Instead, it aligns with the emerging paradigm of precision medicine, emphasizing that personalized therapeutic decisions should be based on individual patient attributes, notably renal function. This approach holds promise for optimizing diuretic therapy, mitigating the frequency of hospital readmissions, and enhancing the overall quality of life for individuals concurrently experiencing AHF and chronic kidney disease (CKD).

One significant challenge in implementing natriuresis-guided therapy is the need for frequent and accurate measurements of urinary sodium excretion. Urine collection and sodium analysis can be cumbersome and may require specialized equipment .

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with acute heart failure (AHF) with reduced ejection fraction either De novo or ADHF.
* Patients with chronic kidney disease (CKD) stages 1-4.
* Patients aged 18 years or older.
* Patients accept to participate in the study.

Exclusion Criteria:

* Patients with significant stenotic valvular diseases (MS, AS).
* Patients with acute coronary syndrome.
* Patients with acute cardiogenic shock.
* Patients with dyspnea primarily due to non-cardiac cause (significant COPD).
* Patients with severe renal impairment requiring dialysis (GFR < 15 mL/min/1.73 m²).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Mean total sodium in urine in both groups. | 24 hours
Duration of the index hospitalization in both groups. | 24 hours

SECONDARY OUTCOMES:
All-cause mortality or HF rehospitalization in both groups. | 90 days
Mean total sodium in urine in both groups. | 90 days
Incidence of arrythmatic complications as AF, VT and incidence of hypokalemia and hypomagnesaemia in both groups. | 90 days
Mean total urine output in both groups. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Salah Eldin Sayed Atta, Supervisor, Study Chair — Assiut University; Heba Mahmoud Abdel-Mohsen El-Naggar, Supervisor, Study Director — Assiut University; Mohamed Abdullah Khalifah, Supervisor, Study Director — South Valley University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Testani JM, Hanberg JS, Cheng S, Rao V, Onyebeke C, Laur O, Kula A, Chen M, Wilson FP, Darlington A, Bellumkonda L, Jacoby D, Tang WH, Parikh CR. Rapid and Highly Accurate Prediction of Poor Loop Diuretic Natriuretic Response in Patients With Heart Failure. Circ Heart Fail. 2016 Jan;9(1):e002370. doi: 10.1161/CIRCHEARTFAILURE.115.002370. PMID 26721915
- [Background] Deferrari G, Cipriani A, La Porta E. Renal dysfunction in cardiovascular diseases and its consequences. J Nephrol. 2021 Feb;34(1):137-153. doi: 10.1007/s40620-020-00842-w. Epub 2020 Sep 1. PMID 32870495
- [Background] Raina R, Nair N, Chakraborty R, Nemer L, Dasgupta R, Varian K. An Update on the Pathophysiology and Treatment of Cardiorenal Syndrome. Cardiol Res. 2020 Apr;11(2):76-88. doi: 10.14740/cr955. Epub 2020 Mar 10. PMID 32256914
- [Background] Brown JR, Uber PA, Mehra MR. The progressive cardiorenal syndrome in heart failure: mechanisms and therapeutic insights. Curr Treat Options Cardiovasc Med. 2008 Aug;10(4):342-8. doi: 10.1007/s11936-008-0054-5. PMID 18647589
- [Background] Oliva-Damaso N, Nunez J, Soler MJ. Spot Urinary Sodium as a Biomarker of Diuretic Response in Acute Heart Failure. J Am Heart Assoc. 2023 Sep 5;12(17):e030044. doi: 10.1161/JAHA.123.030044. Epub 2023 Aug 23. No abstract available. PMID 37609987
- [Background] Martens P, Chen HH, Verbrugge FH, Testani JT, Mullens W, Tang WHW. Assessing intrinsic renal sodium avidity in acute heart failure: implications in predicting and guiding decongestion. Eur J Heart Fail. 2022 Oct;24(10):1978-1987. doi: 10.1002/ejhf.2662. Epub 2022 Sep 6. PMID 36054180
- [Background] Meekers E, Mullens W. Spot Urinary Sodium Measurements: the Future Direction of the Treatment and Follow-up of Patients with Heart Failure. Curr Heart Fail Rep. 2023 Feb;20(1):88-100. doi: 10.1007/s11897-023-00591-4. Epub 2023 Feb 21. PMID 36807114
- [Background] Ter Maaten JM, Beldhuis IE, van der Meer P, Krikken JA, Coster JE, Nieuwland W, van Veldhuisen DJ, Voors AA, Damman K. Natriuresis-guided therapy in acute heart failure: rationale and design of the Pragmatic Urinary Sodium-based treatment algoritHm in Acute Heart Failure (PUSH-AHF) trial. Eur J Heart Fail. 2022 Feb;24(2):385-392. doi: 10.1002/ejhf.2385. Epub 2022 Jan 6. PMID 34791756
- [Background] Ter Maaten JM, Beldhuis IE, van der Meer P, Krikken JA, Postmus D, Coster JE, Nieuwland W, van Veldhuisen DJ, Voors AA, Damman K. Natriuresis-guided diuretic therapy in acute heart failure: a pragmatic randomized trial. Nat Med. 2023 Oct;29(10):2625-2632. doi: 10.1038/s41591-023-02532-z. Epub 2023 Aug 28. PMID 37640861